CLINICAL TRIAL: NCT03331042
Title: A Randomized, Double-Blind, Single-Dose, 4-Way Crossover Study to Assess the Efficacy and Safety of SM-1 (50-mg Diphenhydramine, 5-mg Delayed-Release Zolpidem, and 0.5-mg Delayed-Release Lorazepam) Versus 2 Comparators (50-mg Diphenhydramine and 5-mg Delayed-Release Zolpidem; 50-mg Diphenhydramine and 0.5-mg Delayed-Release Lorazepam) and Placebo in a 5-Hour Phase Advance Model of Transient Insomnia.
Brief Title: SM-1 vs 2 Comparators and Placebo in Participants With a History of Transient Insomnia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sequential Medicine Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SM-A-05
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Transient Insomnia
Keywords: Insomnia; Transient Insomnia; Sleep initiation and maintenance disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): SM-1 (Treatment Period 1), D+Z (Treatment Period 2), D+L (Treatment Period 3), Placebo (Treatment Period 4).
  Interventions: Drug: SM-1; Drug: D+Z; Drug: D+L; Drug: Placebo
- Sequence 2 (Experimental): D+Z (Treatment Period 1), D+L (Treatment Period 2), Placebo (Treatment Period 3), SM-1 (Treatment Period 4).
  Interventions: Drug: SM-1; Drug: D+Z; Drug: D+L; Drug: Placebo
- Sequence 3 (Experimental): D+L (Treatment Period 1), Placebo (Treatment Period 2), SM-1 (Treatment Period 3), D+Z (Treatment Period 4).
  Interventions: Drug: SM-1; Drug: D+Z; Drug: D+L; Drug: Placebo
- Sequence 4 (Experimental): Placebo (Treatment Period 1), SM-1 (Treatment Period 2), D+Z (Treatment Period 3), D+L (Treatment Period 4).
  Interventions: Drug: SM-1; Drug: D+Z; Drug: D+L; Drug: Placebo

INTERVENTIONS:
Drug: SM-1 — 3-drug combination product containing 50-mg diphenhydramine, 5-mg delayed-release zolpidem and 0.5-mg delayed-release lorazepam.
Drug: D+Z — 2-drug combination comparator product containing 50-mg diphenhydramine and 5-mg delayed-release zolpidem.
Drug: D+L — 2-drug combination comparator product containing 50-mg diphenhydramine and 0.5-mg delayed-release lorazepam.
Drug: Placebo — Identical in appearance to SM-1, D+Z and D+L and has the same excipients, but no diphenhydramine, zolpidem, lorazepam or delayed-release coating materials.

SUMMARY:
The purpose of this study is to investigate the effectiveness, safety and tolerability of a combination drug product (SM-1) containing diphenhydramine, zolpidem and lorazepam, in adult participants who sometimes have difficulty in falling asleep or staying asleep, but who do not have chronic insomnia. Participants will receive SM-1, or a combination of diphenhydramine and zolpidem, or a combination of diphenhydramine and lorazepam, or placebo during 4 one-night stays at a sleep center.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent form.
* Experienced at least 1 prior episode of transient insomnia meeting all of the following criteria: difficulty falling asleep or staying asleep; next day impairment or distress associated with the disturbed sleep; frequency of 1 to 7 nights per week; duration of less than 1 month or more than 1 month of intermittent episodes.
* Routinely spends 6.5 - 9.5 hours in bed each night, with bed time varying no more than 2 hours over a week. Potential participants will be required to complete a paper diary for a minimum of 7 days during the screening period, with at least 5 entries completed over the 7 days.
* Body Mass Index (BMI) between 19 and 32 kg/m2.
* Good general health, as determined by a thorough medical, sleep and psychiatric history review, brief physical examination including vital sign measurements, and an assessment of screening laboratory test results.
* Female subjects of childbearing potential must be using an acceptable method of contraception during the study and for the 30 days following the last dose of study drug, and must have a negative urine pregnancy test at every study visit. Female subjects of non-childbearing potential are not required to use contraception if they have been surgically sterilized or are post-menopausal as defined by the cessation of menses for a period of at least 2 years before screening.
* Male subjects must use an acceptable method of contraception during the study and for the 30 days following the last dose of study drug.
* Willing and able to be confined to the study center for 1 night in each of 4 treatment periods, as required by the protocol.
* Refrains from the use of alcohol within 24 hours of check-in for each of 4 treatment periods involving an overnight stay at the study center.
* Refrains from napping (any sleep episode occurring outside subject's main sleep episode) on days of check-in for each of 4 treatment periods involving an overnight stay at the study center.

Exclusion Criteria:

* Females who are pregnant, breast-feeding, or planning a pregnancy during the study period.
* Clinically significant medical disorder or currently unstable medical condition that, in the opinion of the investigator, would confound the results of the study.
* Abnormal laboratory value at screening, judged clinically significant by the investigator.
* History or current evidence of severe hepatic (liver) impairment.
* Clinically significant psychiatric illness, or the history or presence of a major psychiatric illness in the past year.
* Clinically significant abnormal finding on physical examination, as determined by the investigator.
* Lifetime history of seizure disorder (other than childhood febrile seizures) or serious head injury.
* History of chronic insomnia or other sleep disorders, such as sleep apnea, narcolepsy, parasomnia, restless leg syndrome, or circadian rhythm disorder.
* Air travel across more than 2 time zones, an expected change in sleep schedule, or involvement in night work or shift work within 1 month before screening or during the study period.
* Reports a recent history of napping of more than once per week.
* History of alcohol or substance use disorder within the year before screening, or current evidence of alcohol or substance use disorder.
* Self-report of a usual consumption of more than 14 units of alcohol per week. One unit of alcohol is equivalent to 12 ounces of beer, 4 ounces of wine, or 1 ounce of liquor.
* Regular consumption of more than 500 mg of caffeine per day.
* History of routinely smoking during sleep period.
* Discontinuation of smoking or participation in a smoking cessation program within 30 days of screening or plans to discontinue smoking during the study.
* Positive urine drug screen at screening.
* Positive alcohol breathalyzer test at any visit.
* History of allergy or known sensitivity, hypersensitivity, or adverse reaction to diphenhydramine, zolpidem, or lorazepam or other drugs of the same pharmaceutical classes.
* Use of any medication which affects sleep-wake function within 5 half-lives or 2 weeks, whichever is longer, before screening until study completion. This includes prescription, over-the-counter (OTC), and herbal (e.g. valerian root, melatonin) medications.
* Use of any investigational drug within 30 days or 5 half-lives, whichever is longer, before screening.
* Planned surgery (inpatient or outpatient) during the study period.
* Employee or family member of the investigator or study center personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Clinilabs, Inc., New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 22 | 21 | 21 | 21
Completed | 21 | 21 | 20 | 20
Not Completed | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects were randomized to one of four possible planned order of treatments (Sequences) given in the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 22 | 21 | 21 | 21 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (13.68) | 39.3 (13.29) | 36.1 (11.68) | 41.6 (11.77) | 38.9 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 9 | 11 | 43
  Male | 9 | 11 | 12 | 10 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 13 | 10 | 15 | 50
  White | 7 | 6 | 7 | 4 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time (TST)
Description: TST efficacy of SM-1 versus placebo, combination product diphenhydramine plus zolpidem and combination product diphenhydramine plus lorazepam measured by polysomnography (PSG)-defined total sleep time (TST)
Time Frame: 8 hours
Population: Full analysis set consisted of all subjects who were randomized to a treatment sequence, and had taken any study drug.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- SM-1: Subjects received a single dose of the triple drug combination
- Diphenhydramine Plus Zolpidem: Subjects received a single dose of the 2-drug product containing Diphenhydramine plus Zolpidem; i.e., SM-1 without Lorazepam
- Diphenhydramine Plus Lorazepam: Subjects received a single dose of the 2-drug product containing Diphenhydramine plus Lorazepam; i.e., SM-1 without Zolpidem
- Placebo: Subjects received a single dose of a Placebo matching the appearance of the active treatments but containing no active drug components
Arm/Group | SM-1 | Diphenhydramine Plus Zolpidem | Diphenhydramine Plus Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 83 | 83
minutes | 401.82 (68.074) | 404.83 (47.252) | 397.28 (56.982) | 307.38 (107.365)

2. Secondary Outcome: Latency to Persistent Sleep (LPS)
Description: Efficacy of SM-1 versus placebo, combination product diphenhydramine plus zolpidem and combination product diphenhydramine plus lorazepam measured by polysomnography (PSG)-measured sleep induction, the amount of time it takes the subject to fall asleep.
Time Frame: 8 hours
Population: Full analysis set consisted of all subjects who were randomized to a treatment sequence, and had taken any study drug.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- SM-1: Triple drug combination
- Diphenhydramine and Zolpidem: Diphenhydramine and zolpidem
- Diphenhydramine and Lorazepam: diphenhydramine and lorazepam
- Placebo: Placebo
Arm/Group | SM-1 | Diphenhydramine and Zolpidem | Diphenhydramine and Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 83 | 83
minutes | 18.59 (18.548) | 23.10 (29.145) | 23.55 (29.125) | 39.25 (73.961)

3. Secondary Outcome: Number of Awakenings (NAW)
Description: NAW efficacy of SM-1 versus placebo, combination product diphenhydramine plus zolpidem and combination product diphenhydramine plus lorazepam measured by polysomnography (PSG)-measured sleep maintenance.
Time Frame: 8 hours
Population: Full analysis set consisted of all subjects who were randomized to a treatment sequence, and had taken any study drug.
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | SM-1 | Diphenhydramine and Zolpidem | Diphenhydramine and Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 83 | 83
awakenings | 11.0 (6.06) | 10.7 (6.22) | 11.0 (5.91) | 8.6 (5.06)

4. Secondary Outcome: Wakefulness After Sleep Onset (WASO)
Description: WASO efficacy of SM-1 versus placebo, combination product diphenhydramine plus zolpidem and combination product diphenhydramine plus lorazepam measured by polysomnography (PSG)-measured sleep maintenance as the amount of time spent awake after falling asleep.
Time Frame: 8 hours
Population: Full analysis set consisted of all subjects who were randomized to a treatment sequence, and had taken any study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SM-1 | Diphenhydramine and Zolpidem | Diphenhydramine and Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 83 | 83
minutes | 64.11 (66.673) | 58.83 (41.834) | 63.91 (49.841) | 140.06 (99.366)

5. Secondary Outcome: Karolinska Sleepiness Scale (KSS) of Morning Alertness.
Description: Morning alertness measured by Karolinska Sleepiness Scale (KSS). KSS ranges from 1-9, with higher numbers indicating sleepier and lower numbers more alert.
Time Frame: Up to Visit 5
Population: The Safety Population included all subjects that received any study drug, and were grouped by actual treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-1 | Diphenhydramine and Zolpidem | Diphenhydramine and Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 83 | 83
units on a scale | 4.2 (1.99) | 3.9 (2.01) | 3.9 (2.02) | 3.9 (2.01)

6. Secondary Outcome: Number Correct on Digit Symbol Substitution Test (DSST)
Description: Morning alertness measured by DSST. The digit symbol substitution test assesses attention, psychomotor speed, complex scanning, visual tracking, and immediate memory. This test consists of 4 rows each with 25 small blank squares; above each square is a number between 1 and 9. At the top is a 'key,' which pairs each number (1 through 9) with an unfamiliar symbol. The participant has 90 seconds to work as quickly as possible (left to right across the rows) to fill in each blank square with the appropriate symbol based on the number above the square. Results are presented as total number correct; therefore, lower numbers indicate greater impairment. Scores on the DSST range from 0-93
Time Frame: Up to Visit 5
Population: Safety Population included all subjects that received any study drug, and were grouped by actual treatment.
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | SM-1 | Diphenhydramine and Zolpidem | Diphenhydramine and Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 83 | 83
number correct | 56.0 (14.21) | 57.6 (14.98) | 58.3 (16.20) | 60.4 (16.81)

7. Secondary Outcome: Subjective Total Sleep Time (sTST)
Description: Subject reported TST from Post-Sleep Questionnaire (PSQ).
Time Frame: Up to 22 days.
Population: All subjects who were randomized to a treatment sequence, and had taken any study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SM-1 | Diphenhydramine and Zolpidem | Diphenhydramine and Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 82 | 83
minutes | 441.1 (55.97) | 419.0 (79.60) | 422.9 (83.63) | 368.7 (107.47)

8. Secondary Outcome: Subjective Sleep Onset Latency (sSOL)
Description: Subject reported SOL, the amount of time the subject felt it took to fall asleep, from Post-Sleep Questionnaire (PSQ).
Time Frame: Up to 22 days.
Population: All subjects who were randomized to a treatment sequence, and had taken any study drug.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | SM-1 | Diphenhydramine and Zolpidem | Diphenhydramine and Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 82 | 83
minutes | 22.7 (24.30) | 27.7 (34.29) | 26.6 (51.81) | 34.8 (55.53)

9. Secondary Outcome: Subjective Number of Awakenings (sNAW)
Description: Subject reported NAW from Post-Sleep Questionnaire (PSQ).
Time Frame: Up to 22 days.
Population: All subjects who were randomized to a treatment sequence, and had taken any study drug.
Measure: Mean (Standard Deviation); unit: awakenings
Groups:
- Diphenhydramine Plus Zolpidem: Diphenhydramine plus Zolpidem
- Diphenhydramine Plus Lorazepam: Diphenhydramine plus Lorazepam
Arm/Group | SM-1 | Diphenhydramine Plus Zolpidem | Diphenhydramine Plus Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 80 | 82
awakenings | 2.0 (1.73) | 2.2 (2.19) | 2.2 (1.47) | 2.8 (1.83)

10. Secondary Outcome: Number of Participants According to Sleep Quality
Description: Subject reported sleep quality, how well the subject felt he or she slept, from Post-Sleep Questionnaire (PSQ).
Time Frame: Up to 22 days.
Population: All subjects who were randomized to a treatment sequence, and had taken any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-1 | Diphenhydramine and Zolpidem | Diphenhydramine and Lorazepam | Placebo
Number analyzed (Participants) | 84 | 83 | 83 | 83
Participants
  1 = poor | 5 | 3 | 7 | 15
  2 = fair | 13 | 17 | 15 | 39
  3 = good | 43 | 48 | 49 | 21
  4 = excellent | 23 | 15 | 12 | 8

11. Other Pre Specified Outcome: Number of Minutes of Sleep in Stages N1, N2, N3, Rapid Eye Movement (REM) and Latency to REM Onset.
Description: Effect of SM-1 and the two 2-drug combination products (diphenhydramine plus zolpidem and diphenhydramine plus lorazepam) on sleep stage distribution.
Time Frame: 8 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From Day 1 until 7 days after the last dose of study drug.
Arm/Group | SM-1 | Diphenhydramine Plus Zolpidem | Diphenhydramine Plus Lorazepam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/83 | 0/83 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/83 | 0/83 | 0/83
Other Adverse Events (participants affected / at risk) | 3/84 | 2/83 | 1/83 | 1/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SM-1 (N=84) | Diphenhydramine Plus Zolpidem (N=83) | Diphenhydramine Plus Lorazepam (N=83) | Placebo (N=83)
nightmare (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Nightmare
somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — somnolence
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — upper abdominal pain
asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — asthenia
fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — fatigue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT03331042/SAP_000.pdf
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03331042/Prot_001.pdf